CLINICAL TRIAL: NCT02619981
Title: An Objective Assessment of Dental Fear, and the Influence of the Parental Presence on the Behavior of Anxious Children on Their First Restorative Dental Visit
Brief Title: The Effect of Parental Presence on Dental Fear
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr Sharat Pani, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRP/2012/48
Record Dates: First submitted 2015-11-27; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Dental Fear

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Father present (Active Comparator): Child seated at the dental chair, buccal maxillary infiltration anesthesia with 2%Lidocaine administered using a 27 gauge 21mm needle , restorative procedure completed , Father present
  Interventions: Procedure: Restorative procedure; Drug: Maxillary infiltration anesthesia with 2%Lidocaine
- Mother Present (Active Comparator): Child seated at the dental chair, buccal maxillary infiltration anesthesia with 2%Lidocaine administered using a 27 gauge 21mm needle , restorative procedure completed , Mother present
  Interventions: Procedure: Restorative procedure; Drug: Maxillary infiltration anesthesia with 2%Lidocaine
- Both parents present (Active Comparator): Child seated at the dental chair, buccal maxillary infiltration anesthesia with 2%Lidocaine administered using a 27 gauge 21mm needle , restorative procedure completed , both parents present
  Interventions: Procedure: Restorative procedure; Drug: Maxillary infiltration anesthesia with 2%Lidocaine

INTERVENTIONS:
Procedure: Restorative procedure — A restorative dental procedure requiring maxillary buccal infiltration anesthesia, and not exceeding 30 minutes of working time
  Other Names: Dental Filling
Drug: Maxillary infiltration anesthesia with 2%Lidocaine — 1.8ml of 2% Lidocaine with adrenaline administered using a 27 gauge 21mm needle
  Other Names: 2% Lignociane

SUMMARY:
150 children aged between five and seven years presenting for the first dental visit, whose parents consented to participate in the study were selected from patients reporting to the dental clinics Riyadh Colleges of Dentistry and Pharmacy using convenience sampling. Pulse rate for each patient was measured at different clinical situation starting from patient parent separation until end of appointment using a pulse oximeter, Data which collected was statistically analyzed using appropriate statistical analyses using SPSS ver.19 data processing software.

DETAILED DESCRIPTION:
150 children aged between five and seven years presenting for the first dental visit, whose parents consented to participate in the study were selected from patients reporting to the dental clinics Riyadh Colleges of Dentistry and Pharmacy using convenience sampling. Only children who were classified as anxious but able to cope were included in the study (Rating 2 on the Venham's scale).

Pulse rate for each patient was measured at six different clinical situations. 1) Baseline 2) Seating of the child at the chair, 3) Arrival of the dentist, 4) Administration of local anesthesia 5) During the procedure, 6) End of Appointment.

Based on the accompanying person the children were classified as children accompanied by mothers alone, children accompanied by fathers alone, children accompanied by both parents.

The behavior of the child at each situation was recorded using the modified Venham's scale at each interval. The heart rate and oxygen saturation were recorded using pulse oxymetry

ELIGIBILITY:
Inclusion Criteria:

* No previous restorative dental experience
* At least one maxillary posterior tooth requiring restorative care
* Parental consent to participate in the study

Exclusion Criteria:

* Children with previous restorative dental experience
* Children with intellectual disability
* Children with diagnosed neurobehavioral disorders, including (but not limited to ), Autism spectrum disorders, learning disabilities, cerebral palsy, attention deficit hyperactivity disorder

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Child behavior - Subjective | 30min
  Child behavior monitored using the Venham scale

SECONDARY OUTCOMES:
Child Behavior - Objective | 30 min
  Child Behavior Monitored using Pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Hezekiah Mosadomi, DMD, Study Director — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Cox IC, Krikken JB, Veerkamp JS. Influence of parental presence on the child's perception of, and behaviour, during dental treatment. Eur Arch Paediatr Dent. 2011 Aug;12(4):200-4. doi: 10.1007/BF03262807. PMID 21806904
- [Background] Afshar H, Baradaran Nakhjavani Y, Mahmoudi-Gharaei J, Paryab M, Zadhoosh S. The Effect of Parental Presence on the 5 year-Old Children's Anxiety and Cooperative Behavior in the First and Second Dental Visit. Iran J Pediatr. 2011 Jun;21(2):193-200. PMID 23056787
- [Background] Al-Shalan TA, Al-Musa BA, Al-Khamis AM. Parents' attitude towards children's first dental visit in the College of Dentistry, Riyadh, Saudi Arabia. Saudi Med J. 2002 Sep;23(9):1110-4. PMID 12370724
- [Background] Arathi R, Ashwini R. Parental presence in the dental operatory-parent's point of view. J Indian Soc Pedod Prev Dent. 1999 Dec;17(4):150-5. PMID 10863512
- [Background] Marcum BK, Turner C, Courts FJ. Pediatric dentists' attitudes regarding parental presence during dental procedures. Pediatr Dent. 1995 Nov-Dec;17(7):432-6. PMID 8786909